CLINICAL TRIAL: NCT06914830
Title: Musical Video With Virtual Reality Goggles: Effects on Anxiety and Comfort in Ureteroscopic Surgery
Brief Title: The Effect of Musical Video With Virtual Reality Goggles on Patient's Anxiety and Comfort During Ureteroscopy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Hilal Hatice Ülkü, Ass.Prof., Aydin Adnan Menderes University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: musical video show
Record Dates: First submitted 2025-03-21; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Ureteroscopy; Operation Time; Music Listening
Keywords: Ureteroscopy; music therapy; virtual reality; anxiety; comfort
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Following recruitment, patients were divided into study and control groups by randomization (1:1 randomization)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The study group was shown the musical video created by the researchers by taking expert opinions during the surgery.
  Interventions: Other: Musical video demonstration with virtual reality glasses
- Control group (No Intervention): The control group continued to receive the routine care

INTERVENTIONS:
Other: Musical video demonstration with virtual reality glasses — The research was explained to the patient before the operation. The patient was started to watch a video with music with virtual glasses at the 5th minute of the operation and watched it throughout the operation. Two hours after the surgery, the patient who underwent ureteroscopy completed the Data Collection Form, Surgery Specific Anxiety Scale and Perianesthesia Comfort Scale.
  Arms: Experimental group

SUMMARY:
The effect of musical video with virtual reality goggles on patient's anxiety and comfort during ureteroscopy

DETAILED DESCRIPTION:
Ureteroscopy is a surgical procedure used diagnostically or therapeutically in urology. Eliminating the patient's fear, anxiety and worry in the preoperative period is necessary to reduce the surgical stress response seen during the surgical procedure and to ensure normal physiological functions after surgery, early mobilization and patient comfort. When the patient is taken into surgery, reassuring and gentle communication should be established to reduce the patient's anxiety. For this reason, it is important that the surgical team members feel that they are with the patient and make the patient feel that they are with them.

Music is an art that organizes sounds in a way that provides a feeling of happiness. It can help the patient cope with all aspects of the disease; it improves physical, emotional, social and spiritual well-being and can help control and reduce pain and/or agitation. studies examining the relationship between music and depression and anxiety, it was found that depression and anxiety scores were significantly lower in the music therapy group compared to the control group.

The aim of this study was to examine the effect of virtual reality goggles and musical video playback on the patient's operating room anxiety and comfort during ureteroscopy.

The hypotheses that there is no difference in anxiety and comfort levels in the intervention and control groups after music intervention will be tested.

ELIGIBILITY:
Inclusion Criteria:

* Being able to speak and understand Turkish
* Being open to communication
* Being literate
* Being over 18 years of age
* Having a Glasgow Coma Scale score of 13 and above

Exclusion Criteria:

* Visual and hearing impairment
* Previous surgery
* Being a healthcare personnel
* General anesthesia of the patient

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2025-05-10 (Estimated)

PRIMARY OUTCOMES:
Determination of the patient's anxiety levels after the intervention | two hours after surgery
  The Surgery-Specific Anxiety Scale is a five Likert-type scale assessing of anxiety. The reference range of the scale is 0-50, with a higher score reflecting fear of pain, fear of dying during surgery, and fear of postoperative complications and limitations. Cronbach's alpha value of the scale is 0.79.
Determination of the patient's comfort levels after the intervention | two hours after surgery
  The Perianesthesia Comfort Scale is based on a theoretical framework of three levels and four dimensions. It evaluates comfort needs and the achievement of expected comfort improvements. Scale scoring is 24-144 (min-max). Cronbach's alpha: 0.83. A low score indicates poor comfort and a high score indicates good comfort.

CONTACTS AND LOCATIONS:
Overall Officials: Hilal Hatice ÜLKÜ, PhD, Study Chair — Aydin Adnan Menderes University
Locations (1):
- Aydın Adnan Menderes University, Efeler, Aydın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request
Supporting Information: CSR
Time Frame: 6 months after publication
Access Criteria: relevance to the topic of the study and approval of all co-authors within 1 month of receiving the request.